CLINICAL TRIAL: NCT05271019
Title: Efficacy of Early Inspiratory Muscle Training Combined With the Conventional Rehabilitation Programme in Lung Transplanted Patients
Brief Title: Efficacy of Early Inspiratory Muscle Training in Lung Transplanted Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Collaborators: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Laura Muelas Gomez, Clinical physiotherapist, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI 195/21
Record Dates: First submitted 2022-02-16; First posted 2022-03-08 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Lung Transplant Recipients; Muscle Weakness; Respiratory Insufficiency; Pulmonary Rehabilitation; Chronic Lung Disease
Keywords: respiratory muscle training; post lung transplant; breathing exercises; respiratory exercises; pulmonary rehabilitation; exercise capacity
MeSH Terms: conditions — Muscle Weakness; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Investigator, Outcomes Assessor
Masking Description: Neither the professionals in charge of measuring the pre- and post-intervention outcomes nor the statistician are aware of the assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: Conventional Rehabilitation Program (No Intervention): Standard rehabilitation program for 3 months, starting in the early phase in the ICU. A daily session from monday to friday. It includes breathing and secretions management exercises, building upper and lower extremity range of motion. Exercise progression should gradually incorporate aerobic exercises (treadmill, cycloergometer and upper and lower limb strength exercises) and limb strength training.
  Aerobic exercise at moderate intensity (no more than 3-4/10 on the modified Borg scale). Aerobic exercise starting with 20 minutes and gradually increasing up to 30 minutes.
  Limb strength training from 1 to 3 sets of 8-10 repetitions at moderate intensity.
- Experimental group: Conventional Rehabilitation Program + Inspiratory Muscle Training (IMT) (Experimental): Standard rehabilitation program for 3 months, starting in the early phase in the ICU. A daily session from monday to friday. It includes breathing and secretions management exercises, building upper and lower extremity range of motion. Exercise progression should gradually incorporate aerobic exercises (treadmill, cycloergometer and upper and lower limb strength exercises) and limb strength training.
  Aerobic exercise at moderate intensity (no more than 3-4/10 on the modified Borg scale). Aerobic exercise starting with 20 minutes and gradually increasing up to 30 minutes.
  Limb strength training from 1 to 3 sets of 8-10 repetitions at moderate intensity.
  Interventions: Device: Threshold load device

INTERVENTIONS:
Device: Threshold load device — Inspiratory Muscle Training (IMT) for 3 months:
  Though a threshold loading device (5 sets of 6 repetitions, 1session/day, 5 days/week). the inspiratory load will start at 30% of MIP, or up to the maximum patient-tolerable load (max 60% of MIP), no more than 3-5/10 on the modified Borg scale.
  Arms: Experimental group: Conventional Rehabilitation Program + Inspiratory Muscle Training (IMT)

SUMMARY:
Lung transplantation is an effective therapeutic option in the end-stage of chronic respiratory diseases. Lung transplantation improves lung function in terms of capacity and volume. However, the transplanted patient still suffers from muscle weakness and exercise intolerance.

In recent years, respiratory physiotherapy work has intensified in critically ill patients with respiratory muscle weakness and the application of inspiratory muscle training (IMT), which has been shown in several studies to increase inspiratory muscle strength (IMT), improve ventilation and reduce the sensation of shortness of breath. Despite this emerging evidence, inspiratory muscle training (IMT) is not standard practice in most ICUs around the world, nor is it included in a protocolised manner among the components of a pulmonary rehabilitation programme.

Given the limited evidence, the investigators propose to conduct this randomised controlled clinical trial in lung transplant recipients.

The study will compare two groups of transplanted patients, a control group that will follow the rehabilitation programme and standard medical care and another experimental group that will also perform inspiratory muscle training.

This study aims to analyse the effect of IMT on inspiratory muscle strength, exercise capacity and quality of life in lung transplant patients.

DETAILED DESCRIPTION:
For many years, lung transplantation has become an effective therapeutic option for end-stage chronic lung diseases. With transplantation, an improvement in lung function is achieved, achieving volumes and capacities close to those predicted.

After transplantation, muscle deterioration and exercise intolerance are still present; and it will take, according to studies, between 6 months to 1 year to achieve recovery to near normal values. Even in some cases, such as patients with a longer stay in the critical care unit who present a greater deterioration, these values do not reach normal values. In lung transplant recipients, pulmonary rehabilitation including aerobic exercise, resistance exercise and respiratory physiotherapy is the most effective strategy to improve exercise capacity and muscle strength.

Some clinical trials on inspiratory muscle training have identified favourable effects on respiratory muscle fitness and strength.

The purpose of this study is to analyse the impact of early training in lung transplant patients on respiratory muscle strength, exercise tolerance and quality of life. To this end, a randomised controlled trial will be carried out including lung transplant patients (single or double lung adults over 18 years of age) admitted to the hospital where a control group will perform the standard rehabilitation programme: respiratory, aerobic and upper and lower limb strength exercises; while the experimental group will be given inspiratory muscle training with a load of at least 30% of the maximum inspiratory pressure (MIP) in an early manner. Both groups will start the treatment in the critical care unit under conditions of clinical stability (haemodynamic, respiratory and neurologic) and will continue it in hospitalisation. Treatment is performed once a day, 5 days a week from Monday to Friday supervised by a trained physiotherapist.

Every 15 days a data collection will be performed to monitor the follow-up and the data collection will end 3 months after the lung transplantation.

The data collected will be compared from the start of treatment (pre- and post-transplant measurements) and will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Alert or able to cooperate with treatment.
* Able to give Informed Consent and sign it.
* Haemodynamically stable clinical situation or requiring minimal ventilatory support.

Exclusion Criteria:

* Detection of complete paralysis of the diaphragm.
* Progressive neuromuscular diseases or with spinal cord injury.
* Lack of collaboration or cooperation, or non-alertness (Glasgow ≤8).
* Unstable clinical situation (patients requiring high levels of ventilatory support (e.g., Positive End Expiratory Pressure (PEEP)> 10 cmH2O, Fraction Pressure of Inspired Oxygen (FiO2)> 0.60, nitric oxide, nebulised prostacyclin, high frequency oscillation).
* Clinical situation compromising the patient's recovery (cardiac arrhythmias, acute sepsis).
* When the medical treatment team and/or physiotherapy consider that there may be risks.
* Severe pain or dyspnoea that interferes with or impedes the ability to breathe (e.g. rib fracture).
* Patients with lung retransplantation.
* Heart and lung transplant patients.
* When the patient is on palliative treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in respiratory strength: maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) measured in water centimeters (cmH2O). | The groups will be assessed at six times:Pre -Lung transplantation (Pre-LT), at baseline, every 15 days and 3 months after LT
  Maximum respiratory pressure will be measure using a Respiratory Pressure Meter (RPM) named Micro-RPM® . Ever since Black and Hyatt (1969) reported this technique, it is used in healthy control subjects across all ages and athletes. Pressure is recorded at the mouth during quasi-static short (few seconds) maximal breathing according to American Thoracic Society (ATS) guidelines.The maximum value will be obtained. Am J respi Crit Care Med 2002;166:531-535.
Change in functional capacity: 6 minutes walk test (6MWT) measured in meters | The groups will be assessed Pre-LT and 3 months after LT
  6MWT is a submaximal exercise test that entails measurement of distance walked during 6 minutes. The 6MWT provides information regarding functional capacity, response to therapy and prognosis. The test will be in line with American Thoracic Society (ATS) guidelines Statement Guidelines for the Six Minutes Walk Test. Am J respi Crit Care Med 2002;166(1):111-117
Change in Quality of life related with Health(SF-36) measured with a score from 0 to100 | The groups will be assessed Pre-LT and 3 months after LT
  The SF-36 consists of 36 topics that explore eight dimensions of health status: physical function, physical role, bodily pain, general health, vitality, social function, emotional role, and mental health.The SF-36 was previously validated in chronic obstructive pulmonary disease (COPD) patients and has been used in patients before and after lung transplantation (LT). Respiration 2000;67:159-65. Chest 2000;118:408-16.
Change in Respiratory mechanics parameters: respiratory work measured in Joules (J) | The groups will be assessed at baseline, every 15 days and 3 months after LT
  Respiratory mechanics parameters will be analyzed using a POWERbreathe electronic device: the work of breathing is the area for total external inspiratory work as integrated from mouth pressure (cmH2O) and volume (L) signals over time. Physical Therapy 2015;95(9):1264-1273
Change in Inspiratory muscle endurance (Tlim) measure in seconds (s) | The groups will be assessed at baseline, every 15 days and 3 months after LT
  Inspiratory muscle endurance is the time the patient breathe against a submaximal inspiratory load provided by device (POWERbreathe) until task failure due to the symptom limitation. Physical Therapy 2015;95(9):1264-1273.

SECONDARY OUTCOMES:
Changes in dyspnea measured with the modified borg scale 0-10 | The groups will be assessed at baseline, every 15 days and 3 months after LT
  Dyspnea perceptions during the activities of daily living and during exert were assessed. Med Sci Sports Exert 1982; 14: 377-81.
Incidence of atelectasis measured with a score from 0 to 4 | The patients will be assessed through study completion, an average of 3 months
  Registry of Atelectasis is a complete or partial collapse of the whole lung or a part (lobe) of the lung diagnosed by the responsible physician by Chest x-ray report or physician documentation of atelectasis.The postoperative chest radiographs were scored according the following rating (2): 0, no abnormalities; 1, minor atelectasis on one side; 2,minor atelectasis on both sides; 3,major atelectasis on one side; and 4, major atelectasis on both sides. Crit Care Med 2000;28:679-83. Physiotherapy 2011;97(4):278-283
Change in Pulmonary Function measured with Spirometry Test. FEV1/FVC measured in % | The groups will be assessed Pre-LT, at baseline and 3 months after LT
  the investigators will interpret the data obtained from forced spirometry to evaluate how our patient's pulmonary functions is developing after the surgery. FEV1/FVC: It represents the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration (FEV1) to the full, forced vital capacity (FVC).The result of this ratio is expressed as FEV1%. Spirometry is traditionally and widely used to measure pulmonary function and capacity. This test will be performed with a spirometer according to American Thoracic Society (ATS) guidelines and measured in liters . Am J respi Crit Care Med 2002;166:521-522, Eur respi J 2005; 26: 153-161.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Muelas Gómez, PT, MSc, Principal Investigator — Hospital Universitario Puerta de Hierro Majadahonda; Maria de los Angeles Atín Arratibel, MD, PhD, Study Director — Universidad Complutense de Madrid; Maria A Cebria i Iranzo, PT, PhD, Study Director — Hospital Universitario y Politécnico La Fe,Valencia; Ignacio Latorre-Marco, DUE, Study Chair — Hospital Universitario Puerta de Hierro Majadahonda; Montserrat Solis Muñoz, DUE, PhD, Study Chair — Hospital Universitario Puerta de Hierro Majadahonda; Ana Royuela Vicente, Phd, Study Chair — Hospital Universitario Puerta de Hierro Majadahonda; Cristina Ruiz González, PT, Study Chair — Hospital Universitario Puerta de Hierro Majadahonda; Silvia Herguedas Cristobal, PT, Study Chair — Hospital Universitario Puerta de Hierro Majadahonda; Sofia González López, MD, Study Chair — Hospital Universitario Puerta de Hierro Majadahonda
Locations (1):
- Laura Muelas Gómez, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
For now I don't want to share information about the study until I have the protocol or some published results of the intervention. At that time, the information will be shared with the other researchers.

REFERENCES:
- [Background] Pehlivan E, Mutluay F, Balci A, Kilic L. The effects of inspiratory muscle training on exercise capacity, dyspnea and respiratory functions in lung transplantation candidates: a randomized controlled trial. Clin Rehabil. 2018 Oct;32(10):1328-1339. doi: 10.1177/0269215518777560. Epub 2018 May 30. PMID 29843525
- [Background] Nissan Graur PW and MRK. Annals of Physiotherapy Clinics Effects of Inspiratory Muscle Training on Respiratory Muscle Strength , Functional Capacity and Health Related Quality of Life of Patients Following Lung Transplantation. Ann Physiother Clin. 2020;2(1):10-2.
- [Background] Neumannova K, Kuzilkova V, Zurková M, Hubackova L, Michalcikova T, Jakubec P, et al. Respiratory muscle training improves the work of breathing and decreases inspiratory muscle fatigue in patients after lung transplantation. Eur Respir J. 2019 Sep 28;54(suppl 63)
- [Background] Gosselink R, De Vos J, van den Heuvel SP, Segers J, Decramer M, Kwakkel G. Impact of inspiratory muscle training in patients with COPD: what is the evidence? Eur Respir J. 2011 Feb;37(2):416-25. doi: 10.1183/09031936.00031810. PMID 21282809
- [Background] Hoffman M, Augusto VM, Eduardo DS, Silveira BMF, Lemos MD, Parreira VF. Inspiratory muscle training reduces dyspnea during activities of daily living and improves inspiratory muscle function and quality of life in patients with advanced lung disease. Physiother Theory Pract. 2021 Aug;37(8):895-905. doi: 10.1080/09593985.2019.1656314. Epub 2019 Aug 20. PMID 31429627
- [Background] Kendall F, Oliveira J, Peleteiro B, Pinho P, Bastos PT. Inspiratory muscle training is effective to reduce postoperative pulmonary complications and length of hospital stay: a systematic review and meta-analysis. Disabil Rehabil. 2018 Apr;40(8):864-882. doi: 10.1080/09638288.2016.1277396. Epub 2017 Jan 17. PMID 28093920
- [Background] Langer D, Burtin C, Schepers L, Ivanova A, Verleden G, Decramer M, Troosters T, Gosselink R. Exercise training after lung transplantation improves participation in daily activity: a randomized controlled trial. Am J Transplant. 2012 Jun;12(6):1584-92. doi: 10.1111/j.1600-6143.2012.04000.x. Epub 2012 Mar 5. PMID 22390625
- [Background] Candemir I, Ergun P, Kaymaz D, Demir N, Tasdemir F, Sengul F, Egesel N, Yekeler E. The Efficacy of Outpatient Pulmonary Rehabilitation After Bilateral Lung Transplantation. J Cardiopulm Rehabil Prev. 2019 Jul;39(4):E7-E12. doi: 10.1097/HCR.0000000000000391. PMID 31241521
- [Background] Yamaga T, Yamamoto S, Sakai Y, Ichiyama T. Effects of inspiratory muscle training after lung transplantation in children. BMJ Case Rep. 2021 Jul 21;14(7):e241114. doi: 10.1136/bcr-2020-241114. PMID 34290002
- [Background] Langer D, Gosselink R, Pitta F, Burtin C, Verleden G, Dupont L, Decramer M, Troosters T. Physical activity in daily life 1 year after lung transplantation. J Heart Lung Transplant. 2009 Jun;28(6):572-8. doi: 10.1016/j.healun.2009.03.007. Epub 2009 May 5. PMID 19481017